CLINICAL TRIAL: NCT03862118
Title: Evaluation of the Therapeutic Effect of Platelet Rich Plasma (PRP) in Periorbital Hyperpigmentation(POH)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ARYousef, principal investigator, Assiut University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRP in POH
Record Dates: First submitted 2019-03-02; First posted 2019-03-05 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Periorbital Hypermelanosis

STUDY DESIGN:
Intervention Model Description: •The procedure:
  * The face will be washed thoroughly immediately before the procedure.
  * Disinfection with alcohol 70% will be done.
  * A topical anesthetic cream will be applied to the face and left for 30 minutes then it will be removed.
  * The obtained platelet rich plasma will be delivered by intradermal method using mestherapy needle.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PRP — platelet rich plasma will be delivered by intradermal method using mestherapy needle.

SUMMARY:
To evaluate the saftey and efficicacy of autologous PRP in treatment of POH.

DETAILED DESCRIPTION:
Periorbital hyperpigmentation (POH) is a common dermatological condition, also known as periorbital melanosis, periocular hyperpigmentation dark circles under the eyes (DC), infraorbital discoloration, infraorbital darkening, or idiopathic cutaneous hyperchromia of the orbital region. It is a common cosmetic condition that occurs in both sexes and may be considered to be normal variants of pigmentation .

Periorbital hyperpigmentation is a multi-factorial entity.The proposed possible causative factors include genetic or heredity, excessive pigmentation, periorbital edema, thin and translucent lower eyelid skin, venous congestion with hemosiderin deposition, orbital structural problem and shadowing due to skin laxity & tear trough. Other factors such as underlying systemic, metabolic, hormonal diseases, nutritional deficiencies, drugs, allergic reactions, atopic dermatitis, sleep disorders, stress, alcohol consumption, smoking, frequent cosmetic use, frequent eye rubbing and lack of correction for errors of refraction like myopia are also implicated to POH .

Periorbital hyperpigmentation is classified according to Ranu et al into five categories based on the causative factors 1. Constitutional type: seen as typical brownish curved band on lower eyelid or both. 2.Postinflammatory type: irregular patches of brown or grey pigmentation associated with features of lichenification.3. Vascular type: erythema or prominent capillaries or telangiectasia. 4. Shadow effect type: tear trough and eye bags due to sagging skin around eyes. 5. Others: anaemia, hormonal disturbances, nutritional deficiencies and chronic illnesses .

Periorbital hyperpigmentation is graded into four groups according to the severity of the case to be treated;

* Grade1: characterized by faint pigmentation of infraorbital region.
* Grade 2: pigmentation is more pronounced.
* Grade3: deep dark color, all four lids involved.
* Grade 4: grade 3 + pigmentation spreading beyond infraorbital fold .

The diagnosis of POH is mainly clinically, however, a thorough history and clinical assessment is necessary to identify the contributing etiologic factors. The cutaneous examination should be evaluated to detect the involvement of eyelids, extend beyond the periorbital region, color of hyperpigmentation, presence of any dermatological disease or scar, presence of any visible bulging, skin laxity, tear trough, superficial visible vasculature, in infraorbital region presence of pigmentation in other areas .

Eye lid stretch test or manual stretching of the lower eyelid skin can help to differentiate between true pigmentation and shadowing effect .

Wood's lamp examination is done to differentiate between the epidermal and dermal pigmentation.The variations in epidermal pigmentation become more apparent under Wood's light. For dermal pigmentation, this contrast is less pronounced .

Dermatoscopy: It is a non-invasive diagnostic technique for the in vivo observation of pigmented skin lesion allowing a better visualization of surface and subsurface structures and being easy and feasible to use. It can be used to differentiate the type of POH whenever there is doubt while examining with naked eyes. The dermatoscopic findings of POH are- a) Vascular type: diffuse erythema pattern or multiple thin blood vessels or diffuse vascular network, b) Pigmented type: a pattern of multiple dots with different sizes and colors or a diff use network of pigments and c) Mixed type: Combination of vascular and pigmented type .

Treatment of POH:

There are a number of treatment options available for POH. Among the available treatment options for POH include:

1. Topical Applications: The various topical bleaching agents are hydroquinone, kojic acid, a triple combination, azelaic acid, arbutin, topical vitamin C. Out of these topical agents the most widely used is hydroquinone, used in a strength of 2% to 6% .
2. Chemical Peelings: Chemical peelings could be used alone or in combination therapy with topical treatments. Glycolic acid 20% is the most commonly used peeling in the treatment of POH. Lactic acid 15% + TCA 3.75% combination is very effective treatment option for POH .
3. Lasers: lasers have been used increasingly in cosmetic dermatology. Periorbital hyperpigmentation has been successfully treated with various noninvasive lasers that target pigment and vascularity. Various lasers that have been used for treating dark circles are: Q switched ruby laser (694 nm), Q switched alexanderite laser, and Nd:Yag laser (1064nm).
4. Platelet-rich plasma (PRP): PRP is a generic term used to describe a plasma suspension obtained from whole blood, prepared so as to contain platelet concentrations higher than those normally found in circulating blood.

The mechanism of action of PRP is based on the fact that platelets contain many growth factors in their alpha granules. These factors have a well-known role in the process of tissue repair. Thus, the concentration of these substances in injured tissues could be beneficial to providing more agility to the regeneration processes .

PRP treatment is mainly effective for wrinkles, laxity, and secondary PIH-related dark circles. PRP can stimulate dermal fibroblast proliferation and collagen synthesis (Kim DH et al, 2011). Transforming growth factor-β1 and epidermal growth factor in PRP are suggested to inhibit melanin production via delayed extracellular signal-regulated kinase activation and inhibition of prostagandin-E2 expression/ tyrosinase enzyme activity, respectively (Yun WJ et al, 2013). In addition, PRP improves fat graft survival and can be used in combination with autologous fat grafts for dark circles

ELIGIBILITY:
Inclusion Criteria:

* •Both sexes will be included.

  * Age (20-50)
  * Patient with Fitzpatrick skin types III-IV

Exclusion Criteria:

* • Patients with known platelet dysfunction syndrome, critical thrombocytopenia (<50,000/ul), any hemodynamic instability.

  * Patients with chronic medical illness (e.g. diabetes, chronic infections, and blood dyscrasias).
  * Patients with local inflammatory skin disorders or active herpes infection at the site of the procedure.
  * Patients on consistent use of anti-coagulants or non-steroidal anti-inflammatory drugs (NSAID) within 48 hours of procedure.
  * Haemoglobin level< 10 g/dl were also excluded.
  * Patients with cancer- especially hematopoietic or of bone.
  * Pregnant females.
  * Patients with corticosteroids injection at treatment site within 1 month or systemic use of corticosteroids within 2 weeks.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
cure rate | 6 months
  assess cure rate of PRP in treatment of POH

CONTACTS AND LOCATIONS:
Overall Officials: azza rady, doctor, Principal Investigator — Assuit university hospital

REFERENCES:
- [Derived] Badran AY, Abd Elazim NE, Yousef AR, Mekkawy MM. Platelet-Rich Plasma Injections in Periorbital Hyperpigmentation in Skin Phototypes III and IV: Strengthening the Assessment of Treatment Outcomes. Dermatol Surg. 2025 Jan 1;51(1):61-66. doi: 10.1097/DSS.0000000000004372. Epub 2024 Aug 20. PMID 39163646